CLINICAL TRIAL: NCT01220596
Title: A Randomized, Multi Center, Phase IIIb Open-label Study to Evaluate the Efficacy of Sequential Therapy of Peginterferon Alfa-2a(Pegasys(TM)) Following Entercavir Compared With Peginterferon Alfa-2a Monotherapy in Patient With HBeAg Positive Chronic Hepatitis B.
Brief Title: Efficacy Study of Sequential Therapy of Peginterferon Alfa-2a Following Entecavir in Patient With Chronic Hepatitis B.
Acronym: POTENT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Joo Hyun Sohn / Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25206
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential therapy (Experimental): Entecavir/Baraclude(TM), 0.5mg, oral administration, once daily, for the first 12 weeks Pegylated interferon α-2a/Pegasys(TM), 180mcg, subcutaneous injection. once a week, from week 4 to 52 for 48 weeks
  Interventions: Drug: Entecavir and Pegylated interferon α-2a Sequential Treatment Group
- Peginterferon alfa-2a monotherapy (Active Comparator): Pegylated interferon α-2a/Pegasys(TM), 180mcg, subcutaneous injection. once a week, for the first 48 weeks
  Interventions: Drug: Pegylated interferon α-2a Monotreatment Group

INTERVENTIONS:
Drug: Entecavir and Pegylated interferon α-2a Sequential Treatment Group — Entecavir/Baraclude(TM), 0.5mg, oral administration, once daily, for the first 12 weeks Pegylated interferon α-2a/Pegasys(TM), 180mcg, subcutaneous injection. once a week, from week 4 to 52 for 48 weeks
  Other Names: Generic/Brand name: Pegylated interferon α-2a/Pegasys(TM); Generic/Brand name: Entecavir/Baraclude(TM)
  Arms: Sequential therapy
Drug: Pegylated interferon α-2a Monotreatment Group — Pegylated interferon α-2a/Pegasys(TM), 180mcg, subcutaneous injection. once a week, for the first 48 weeks
  Other Names: Generic/Brand name: Pegylated interferon α-2a/Pegasys(TM)
  Arms: Peginterferon alfa-2a monotherapy

SUMMARY:
Evaluate the safety and efficacy of Peginterferon alfa-2a following Entecavir compared with Peginterferon alfa-2a monotherapy in patient with HBeAg positive chronic hepatitis B.

* Increased HBeAg seroconversion rate
* Increased HBsAg loss rate
* To define the best treatment condition for chronic HBV hepatitis patients

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B patients with HBeAg positive, HBsAg positive, HBV DNA > 100,000 copies/ml and anti-HBs negative, serum ALT exceeding 2 X ULN but less than 10 X ULN.

Exclusion Criteria:

* Patient infected concurrently with HCV, HDV and HIV or patient with a history of antiviral treatment for Hepatitis B or patient with hepatic decompensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
HBeAg seroconversion | 24 weeks after treatment

SECONDARY OUTCOMES:
the change of HBsAg titer | 24 weeks after treatment
the rate of combined HBeAg seroconversion and HBV DNA < 300 copies/ml | 24 weeks after treatment
The rate of serum HBV DNA < 300 copies | 24 weeks after treatment
The rate of ALT normalization | 24 weeks after treatment
The rate of HBsAg loss | 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joo Hyun Sohn, MD, Ph.D, Principal Investigator — Hanyang University
Locations (20):
- South Korea (20):
  - Dong-A University Medical Center, Busan, Busan
  - Kosin University Gospel Hospital, Busan, Busan
  - Inje University Haeundae Paik Hospital, Busan, Busan
  - Dankook University Hospital, Cheonan, Chungcheongnam-do
  - Kyungpook National University Hospital, Daegu, Daegu
  - Yeungnam University Medical Center, Daegu, Daegu
  - Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Bundang CHA medical center, Sungnam, Gyeonggi-do
  - Busan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeju National University Hospital, Jeju City, Jeju-do
  - Kangbuk Samsung Hospital, Seoul, Seoul
  - Kyunghee university Medical Center, Seoul, Seoul
  - Hanyang University Hospital, Seoul, Seoul
  - Kangdong Sacred Heart Hospital, Seoul, Seoul
  - Kangnam Severance Hospital, Seoul, Seoul
  - Inje University Sanggye Paik Hospital, Seoul, Seoul
  - Konkuk University Medical Center, Seoul, Seoul

REFERENCES:
- [Derived] Jun DW, Ahn SB, Kim TY, Sohn JH, Kim SG, Lee SW, Kim BH, Kim DJ, Kim JK, Kim HS, Hwang SG, Choi WC, Tak WY, Lee HJ, Yoon KT, Yun BC, Lee SW, Baik SK, Park SH, Park JW, Park SJ, Lee JS. Efficacy of Pegylated Interferon Monotherapy versus Sequential Therapy of Entecavir and Pegylated Interferon in Hepatitis B e Antigen-Positive Hepatitis B Patients: A Randomized, Multicenter, Phase IIIb Open-Label Study (POTENT Study). Chin Med J (Engl). 2018 Jul 20;131(14):1645-1651. doi: 10.4103/0366-6999.235880. PMID 29998882